CLINICAL TRIAL: NCT06876740
Title: Project Safe Guard-Trauma (PSG-T): A Randomized Controlled Trial of Counseling to Promote a Secure Home Environment
Brief Title: Project Safe Guard-Trauma
Acronym: PSG-T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-1287; HT9425-24-1-0693 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: PTSD; Firearm Injury; Suicide Prevention; Firearm Safety
Keywords: PTSD; Firearm Injury; Suicide Prevention; Firearm safety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Participants who meet inclusion and exclusion criteria will be equally randomized between the two intervention conditions following the pre-intervention assessment. We will use computerized block randomization to allocate participants into either Project Safe Guard-Trauma or Project Safe Guard. Block randomization will vary by the number of participants in each block to ensure that the research staff cannot anticipate the next randomization, thereby reducing potential for bias. Biostatisticians will oversee randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project Safe Guard - Trauma (Experimental): Participants randomized into this arm will be offered Project Safe Guard-Trauma (PSG-T), which is a brief, single-session intervention designed to promote secure firearm storage practices among individuals with PTSD. Participants in this arm will also receive crisis response planning (CRP).
  Interventions: Behavioral: Project Safe Guard - Trauma
- Project Safe Guard (Active Comparator): Participants randomized into this arm will be offered Project Safe Guard (PSG), which is a brief, single-session intervention designed to promote secure firearm storage practices. Participants in this arm will also receive crisis response planning (CRP).
  Interventions: Behavioral: Project Safe Guard

INTERVENTIONS:
Behavioral: Project Safe Guard - Trauma — Project Safe Guard-Trauma (PSG-T) is a brief (15- to 20-minute), single-session lethal means safety counseling intervention (LMSC) for firearm-owning individuals with posttraumatic stress disorder (PTSD). PSG-T is designed to promote secure firearm storage practices by (1) using motivational interviewing techniques and (2) addressing the functional link between PTSD symptoms and unsafe firearm storage practices. In motivational interviewing-based LMSC, the clinician uses a guided approach to help individuals identify their values and motivations for secure firearm storage, rather than prescribing a certain set of actions. The focus is on respecting patients' autonomy and normalizing responsible firearm ownership by developing discrepancies, amplifying ambivalence, expressing empathy, rolling with resistance, and supporting self-efficacy. PSG-T combines PSG-proven motivational interviewing techniques with PTSD- and firearm-specific psychoeducation.
  Arms: Project Safe Guard - Trauma
Behavioral: Project Safe Guard — Project Safe Guard-Trauma (PSG) is a brief (15- to 20-minute), single-session lethal means safety counseling intervention (LMSC) for firearm-owning individuals. PSG-T is designed to promote secure firearm storage practices by using motivational interviewing techniques. In motivational interviewing-based LMSC, the clinician uses a guided approach to help individuals identify their values and motivations for secure firearm storage, rather than prescribing a certain set of actions. The focus is on respecting patients' autonomy and normalizing responsible firearm ownership by developing discrepancies, amplifying ambivalence, expressing empathy, rolling with resistance, and supporting self-efficacy.
  Arms: Project Safe Guard

SUMMARY:
The goal of this randomized controlled trial is to determine if a counseling intervention, Project Safe Guard-Trauma (PSG-T), increases secure firearm storage practices in adults who screen positive for posttraumatic stress disorder (PTSD). The main questions this study aims to answer are:

* Does PSG-T lead to more secure firearm storage practices?
* Does PSG-T increase knowledge about the link between firearm storage practices and suicide risk?
* Does PSG-T increase intentions to store firearms securely?

Researchers will compare PSG-T to a control, Project Safe Guard (PSG), which is a counseling intervention that does not focus on the potential influence of PTSD symptoms on firearm storage practices. This will help to determine if PSG-T works better than PSG to increase secure firearm storage in adults with elevated PTSD symptoms.

Participants will:

* Complete a baseline survey
* Receive the counseling intervention
* Complete a survey immediately after the intervention and at 1-, 3-, and 6-months following the intervention

DETAILED DESCRIPTION:
Firearms are the most common suicide method among service members, veterans, and civilians. Secure firearm storage reduces the risk of suicide. Lethal means safety counseling (LMSC) is an effective approach to promote secure firearm storage and, therefore, decrease the risk of suicide. Suicide risk is elevated among individuals with posttraumatic stress disorder (PTSD). PTSD affects safety perceptions and firearm storage practices. Current data indicate that the gold standard existing LMSC intervention - Project Safe Guard (PSG) - has reduced efficacy for individuals with elevated PTSD symptoms. Thus, there is a need to adapt LMSC for individuals with elevated PTSD symptoms.

Project Safe Guard-Trauma (PSG-T) is a brief LMSC intervention rooted in PSG principles but adapted specifically for firearm-owning individuals with PTSD. This study will evaluate the efficacy of PSG-T compared with control (standard PSG) in prompting more secure firearm storage behaviors. This study is a 2-arm randomized controlled trial. Participants will be randomized following the pre-intervention assessment. The participants will receive a single-session LMSC intervention, post-intervention assessment, and 1-, 3-, and 6- month follow-up assessments. The goal is to increase knowledge about the link between firearm storage practices and suicide risk, intentions to store firearms safely, and actual safer firearm storage behaviors.

Aim 1: To conduct a 2-armed randomized control trial to evaluate the efficacy of PSG-T compared with a control (PSG) in increasing knowledge about the link between firearm storage practices and suicide risk, intentions to store firearms safely, and actual safer firearm storage behaviors.

Hypothesis 1: Compared with PSG, at 1-, 3-, and 6-month follow-up, PSG-T will result in greater (a) knowledge about the link between firearm storage practices and suicide risk, (b) intentions to store firearms securely, and (c) actual more secure firearm storage behaviors (primary outcome at 6-month follow-up).

Aim 2: To evaluate differences in PTSD-related negative cognitions about the world as a potential mechanism of change in PSG-T for increasing knowledge, intentions, and behaviors regarding safe firearm storage practices.

Hypothesis 2: Participants who receive PSG-T will report fewer PTSD-related negative cognitions about the world compared with participants who receive PSG, and these decreases will be associated with increases in (a) knowledge about the link between firearm storage practices and suicide risk, (b) intentions to store firearms securely, and (c) actual more secure firearm storage behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+ years
* Firearm owner
* History of one or more victimization traumas per the Life Events Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) (LEC-5), defined as having directly experienced physical assault, sexual assault, combat, and/or captivity
* Positive posttraumatic stress disorder (PTSD) screen on the Primary Care PTSD Screen for DSM-5 (PC-PTSD-5)
* Willing to provide physical location at time of Zoom sessions
* Willing to keep Zoom camera on during study sessions
* Ability to read, write, and speak English

Exclusion Criteria:

* Currently stores all personal firearms unloaded and locked
* Active psychosis or acute mania necessitating clinical intervention
* Acute thoughts of self- or other-harm necessitating imminent clinical intervention (e.g., hospitalization)
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2028-06-14 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Firearm Storage Practices | Baseline to 6-Month Follow-Up
  The primary endpoint is the improvement in actual secure firearm storage practices, as measured at the 6-month follow-up assessment, compared with baseline. The firearm storage assessment includes a grid question asking whether personally owned firearms are locked or unloaded-indicating secure storage practices. Participants can indicate that "none," "some," or "all" of their firearms are in an unloaded or locked condition.
  We assign a score of 2 if the secure practice applies to all firearms, 1 if it applies to some firearms, and 0 if it applies to none. A higher score corresponds to more secure storage practices. The maximum score, achieved when all firearms are both unloaded and locked, is 4, while the minimum score is 0. Improvement will be defined as a change score > 0 between the pre-intervention and 6-month follow-up assessments.

SECONDARY OUTCOMES:
Knowledge of Firearm Storage Practices and Suicide Risk Link | Baseline to 6-Month Follow-Up
  Participants will be asked, "To what extent do you think owning a firearm is related to suicide risk?" and "To what extent do you think how a firearm is stored (e.g., unlocked, loaded) is related to suicide risk?" Responses are captured on a 5-point Likert scale (1 = Not at all, 2= Slightly, 3 = Moderately, 4 = Strongly, 5 = Extremely).
Intentions to Securely Store Firearms | Baseline to 6-Month Follow-Up
  Participants will be asked: (a) "How likely would you be to adhere to your clinician's recommendations to store your firearm locked for safety purposes?" and (b) "How likely would you be to adhere to your clinician's recommendations to store your firearm unloaded for safety purposes?" Responses are captured on a 5-point scale (1 = Very Unlikely, 2 = Unlikely, 3 = Neutral/Possibly, 4 = Likely, 5 = Very Likely).
Posttraumatic Cognitions Inventory (PTCI) negative-world subscale | Baseline to 6-Month Follow-Up
  Posttraumatic stress disorder-related negative cognitions about the world will be evaluated using the Posttraumatic Cognitions Inventory (PTCI). The PTCI is a 33-item self-report measure of negative cognitions about the self and world and self-blame. Respondents rate the degree to which they agree or disagree with each statement on a 7-point scale (1 = Totally disagree, 2 = Disagree very much, 3 = Disagree slightly, 4 = Neither agree nor disagree, 5 = Agree slightly, 6 = Agree very much, 7 = Totally agree). We will use the total score of the 7-item PTCI negative-world subscale to measure the purported mediator of change of Project Safe Guard-Trauma
Client Satisfaction Questionnaire-8 (CSQ-8) | Baseline to 6-Month Follow-Up
  Participant acceptability of services will be evaluated using the Client Satisfaction Questionnaire-8 (CSQ-8), an 8-item self-report measure. Each item evaluated using varying descriptive scales with corresponding numerical values. Scores are summed across items, with higher values indicating greater acceptability of the services received.
Posttraumatic Stress Disorder (PTSD) Checklist for Diagnostic and Statistical Manual of Mental Illness-5 (DSM-5) (PCL-5): | Baseline to 6-Month Follow-Up
  PTSD symptoms will be evaluated using the PTSD Checklist for DSM-5 (PCL-5), a 20-item self-report measure. Participants rate the severity of each symptom over the past month on a 5-point scale (0 =Not at all, 1 = A little bit, 2 = Moderately, 3 = Quite a bit, 4 = Extremely). A composite score is generated from responses with symptom cluster scores corresponding to DSM-5 diagnostic criteria (i.e., intrusions, avoidance, negative alterations in cognitions and mood, hyperarousal); higher scores reflect more severe PTSD symptomatology.
Depressive Symptom Index-Suicidality Subscale (DSI-SS) | Baseline to 6-Month Follow-Up
  Suicidal ideation severity over the past 2 weeks will be evaluated using the Depressive Symptom Index-Suicidality Subscale (DSI-SS), a 4-item self-report measure. Respondents rate each item on a 4-point scale ranging from 0 to 3 (e.g., Item 1: 0 = I do not have thoughts of killing myself; 1 = Sometimes I have thoughts of killing myself; 2 = Most of the time I have thoughts of killing myself; 3 = I always have thoughts of killing myself). A total score ranging from 0 to 12 is calculated from summed responses, with higher scores indicating more severe suicidal ideation.
Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R) | Baseline to 6-Month Follow-Up
  The self-report SITBI-R assesses various aspects of self-injurious thoughts and behaviors. The evaluation measures will only include the questions about the lifetime occurrence of the target construct (e.g., the suicidal ideation module asks respondents, "Have you ever had thoughts of killing yourself?").

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
This trial involves sensitive participant information, including information regarding suicidality, mental health, and firearm ownership and requires careful handling to prevent any negative impact on participants or their families.

REFERENCES:
- See also: University of Colorado Anschutz Medical Campus Department of Emergency Medicine Funded Research — https://medschool.cuanschutz.edu/emergency-medicine/research/funded-research